PRINCIPAL INVESTIGATOR: Robert J. Kreitman, M.D.

**STUDY TITLE:** Randomized Phase II Trial of Rituximab with Either Pentostatin or

Bendamustine for Multiply Relapsed or Refractory Hairy Cell Leukemia

**STUDY SITE:** NIH Clinical Center

Cohort: *Affected patients* 

Consent Version: 09/21/2022

#### WHO DO YOU CONTACT ABOUT THIS STUDY?

**Study PI:** Robert J. Kreitman, M.D

Phone: 301-480-6187

Email: kreitmar@mail.nih.gov

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

The remaining document will now describe the research study in more detail. This information should be considered before you make your choice. Members of the study team will talk with you about the information described in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research interventions in which they would want to participate. Take the time you need to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers.

If the individual being asked to participate in this research study is not able to give consent to be in this study, you are being asked to give permission for this person as their decision-maker. The term "you" refers to you as the decision-maker and/or the individual being asked to participate in this research, throughout the remainder of this document.

## IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

#### WHY IS THIS STUDY BEING DONE?

To see how effective the treatment for hairy cell leukemia (HCL) or HCL variant (HCLv) is using pentostatin plus rituximab or bendamustine plus rituximab. There has never been a study to compare which combination of treatments works best for HCL/HCLv.

## Why are you being asked to take part in this study?

You have HCL or HCLv and you are in need of treatment.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)

Version Date: 09/21/2022


## How many people will take part in this study?

This study plans to enroll up to 72 patients.

This is a randomized study of pentostatin plus rituximab versus bendamustine plus rituximab for multiply relapsed HCL and HCLv. The primary objective of the study is to determine if response in each regimen is higher than what you might expect from rituximab alone, and to determine which regimen might be better. Before the protocol begins to randomize the patients, it will be necessary to make sure the proposed dose of bendamustine plus rituximab, which has been shown to be safe in a similar form of leukemia, is also well tolerated in HCL/HCLv. 12 patients will therefore receive bendamustine plus rituximab without being randomized. If toxicity is observed in HCL/HCLv patients, which is more than what we would expect from other leukemia patients, the protocol may need to be changed before patients get randomized. Otherwise, the optimal bendamustine-rituximab dose will be considered appropriate and patients will then be randomized to receive either this dose of bendamustine + rituximab, or pentostatin plus rituximab. If you take one treatment, and either get worse or respond but then relapse, you may then 'cross over' to the other regimen, as long as you are still eligible. If you previously received one of the regimens and did not respond, you may receive the other regimen only and you would not be in the groups that would be compared.

# **Description of Research Study**

This consent form is for the treatment of hairy cell leukemia (HCL) and HCL variant with pentostatin and rituximab or bendamustine plus rituximab. Another name for rituximab is Rituxan. Rituximab is a monoclonal antibody which binds to the hairy cells and may kill them either by causing the cells to kill themselves, or by getting the immune system to kill the cells. Rituximab is also effective in HCL but is not considered standard treatment and it has not been used as long as cladribine or pentostatin for this disease. Antibodies are proteins that can protect the body from foreign invaders, such as bacteria and viruses, by binding to substances called antigens. Rituximab works by binding to a protein, called the CD20 protein (which is found on the surface of normal and cancerous B-lymphocytes), which helps to destroy the B-lymphocytes. It is given intravenously (through a vein) over a period of several hours. Rituximab has been approved by the Food and Drug Administration (FDA) for several forms of leukemia, lymphoma and rheumatoid arthritis. Bendamustine is a chemotherapy drug which is given intravenously.

Bendamustine is approved for chronic Lymphocytic leukemia (CLL) and non-Hodgkin's lymphoma. Its use in HCL/HCLv has not been reported.

Pentostatin is a chemotherapy drug which has been used for HCL for over 20 years and is approved for HCL. It is given by an intravenous injection or diluted in a larger volume and given over 20 to 30 minutes. The combination of pentostatin and rituximab has been reported to have been used in 7 patients with HCL, and is effective, but no single trial treating patients with this combination has been reported.

Whether you receive pentostatin plus rituximab or bendamustine plus rituximab is not up to you, but is determined in a random way which you and your doctors cannot control. It is like the flip of a coin. If you are among the first 12 patients in the study you will receive bendamustine plus rituximab. The rituximab is given over about 2 hours, although it may be given more slowly if

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


needed, especially the first few times. Rituximab and pentostatin are given every 2 weeks for a total of 12 doses of each.

Bendamustine is given over 30 to 60 minutes on the 1<sup>st</sup> and 2<sup>nd</sup> days of cycles 4 weeks apart. Patients would receive 6 cycles. On these 4-week cycles, rituximab is given every other week for 12 doses, just like patients receiving pentostatin and rituximab. It is not known whether one drug combination with rituximab is better than the other. This research trial allows you to receive up to 24 infusions of rituximab, and if you are benefiting and require more treatment, you may be referred back to your referring doctor for the additional treatment. As part of this study, you will have many lab tests, including bone marrow biopsies and blood tests, to determine whether you have hairy cells left during or after treatment. This protocol will allow lab tests to be performed either at NIH or by your local physician.

## What will happen if you take part in this research study?

## Before you begin the study therapy

You were already found to be eligible for this study. Before you begin study therapy, you will have several tests performed to confirm that the study is suitable for you. Your doctor will review your medical history and the drugs that you are currently taking as well as the previous treatments of your disease to confirm whether you can participate in this study.

Some of these tests or procedures are part of regular care and may be done even if you are not being considered to join the study. If you have had some of these tests or procedures recently, they may or may not have to be repeated. The following tests and procedures will be performed prior to starting treatment:

You will also have additional samples collected for research tests. Up to ½ cup of blood may be collected at each visit.

- Lab blood and urine tests will be collected to check your health. Other blood samples will be collected for research
- Electrocardiogram (EKG) of the heart will be done to check the electrical activity of your heart
- Echocardiogram of the heart will be done to check how well your heart pumps.
- Stress test to check how your heart works during physical activity
- Test to evaluate how well your lungs work
- CT scan and/or MRI (with or without contrast)
- Abdominal ultrasound to check the major organs in the abdominal cavity

## **During the study**

- History and physical exam to check your health
- Electrocardiogram (ECG)

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


Page **3** of **18** 

- Tumor measurements will be obtained from the computed tomography or CT scan of your neck, chest, abdomen, and pelvis and/or MRI. Many patients will undergo ultrasound tests instead of CTs
- Routine blood and urine tests and research blood to determine amount of hairy cells in your blood.
- Bone Marrow biopsy with aspirate, blood flow cytometry, Spine MRI, and CT or ultrasound at:
  - Prior to cycle 4
  - 4-6 weeks after your counts (CBC) show you are in complete remission
  - Yearly while in complete remission for 4 years
  - Every 2 years thereafter while in complete remission

## **Study Chart:**

#### **Randomization and Initial**

#### **Treatment:**

| | Cycles<br>1-6 | | |
|--------------|---------------|----|-----|
| Study | d1 | d2 | d15 |
| Treatment | | | |
| Bendamustine | X | X | |
| Pentostatin | X | | X |
| Rituximab | X | | X |

<sup>\*</sup>cycles will repeat every 28 days (+/- 2 days)

#### **Birth Control**

If you are breast feeding or pregnant, you may not take part in the study because we don't know how this medicine would affect your baby or your unborn child. If you are able to become pregnant, or are the partner of someone who can become pregnant, you will need to practice an effective form of birth control before starting study treatment, during study treatment, and for 12 months after you finish study treatment. If you think that you or your partner is pregnant, you should tell your study doctor or nurse at once.

Effective forms of birth control include

- Abstinence
- intrauterine device (IUD)
- hormonal [birth control pills, injections, or implants]
- tubal ligation
- vasectomy

## PATIENT IDENTIFICATION | Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


## **Risks or Discomforts of Participation**

## What side effects or risks can I expect from being in this study?

#### Rituximab toxicity

Rituximab is generally well tolerated by most patients. However, it can cause side effects. You may have none, some, or all of the effects listed below, and they may be mild, moderate, or severe. In some instances, patients who have used rituximab have died. You will be closely monitored by medically trained staff for any side effects and should report any changes in the way you feel to your study doctor. Some side effects may require treatment with medications, procedures, or other therapies. If you develop certain side effects, you may need a break from taking rituximab. Many side effects will improve or go away; however, some can be long lasting or permanent. If you have questions about the risks of rituximab please talk to your study doctor.

## Likely (50-60% of patients):

Fever

## Less likely (25-50% of patients):

- Decrease in lymphocyte type of normal white blood cells
- Chills
- Infection
- Fatigue

## Unlikely (10-25% of patients):

- Nausea
- Headache
- Night Sweats
- Rash
- Abdominal pain
- Decrease in normal white blood cells
- Decrease in neutrophil type of normal white blood cells (neutrophils are cells which help fight infection)
- Itching
- Increased cough,
- Low platelets (cells which help blood clotting)
- Runny nose
- Back pain
- Low blood pressure
- Diarrhea
- Vomiting
- Muscle pains
- Joint pains
- Dizziness

**Infusion-Related Reactions** - Rituximab may cause side effects associated with infusion of the drug through the veins. Such side effects are called infusion related reactions. Infusion-related

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


reactions can occur up to 24 hours after receiving rituximab, but they usually happen within 30 minutes to 2 hours of beginning an infusion. Most infusion-related reactions are mild or moderate in severity, but they can be severe, and may even lead to death. Most reactions occur with the first infusion and improve with later infusions. Data indicate that symptoms of an infusion-related reaction occur in about 77% of people after their first dose of rituximab (severe symptoms occur in about 7%). By the eighth dose, the rate of such symptoms decreases to approximately 14%. The most common symptoms include fever, chills, nausea, dizziness, vomiting, headache, sweating, flushing, itching, skin rash, hives, runny nose, sneezing, cough, fatigue, joint pain, muscle pain, swelling of arms or legs, soreness or swelling at disease sites, and chest pain. Severe reactions may include tongue or throat swelling, wheezing or difficulty breathing, fluid or inflammation in the lungs, low blood pressure, irregular heartbeat, and heart attack. Notify your doctor immediately if you experience any of the symptoms above while receiving, or soon after receiving, an infusion of rituximab.

**Tumor Lysis Syndrome** – Some patients can develop tumor lysis syndrome after rituximab treatment. Tumor lysis syndrome is caused when cancer cells break down and release their contents into your blood. Tumor lysis syndrome can lead to high levels of potassium in the blood, changes in the blood levels of other electrolytes, kidney failure, and can cause death in severe cases.

**Skin and Mucous Membrane Reactions** – Reactions of the skin and/or mucous membranes (the lining of the mouth, nose and eyes) may occur with rituximab. Examples of this type of reaction include peeling, rashes, blisters, and open sores. While these reactions appear to be rare, they can be severe or even lead to death when they occur. They usually occur from 1 to 13 weeks after receiving rituximab. If you experience any of these symptoms, contact your study doctor immediately.

**Infections** - Rituximab may increase your risk of developing certain types of infections. Some of these infections can be serious or lead to death. It is important to tell your doctor immediately if you develop symptoms of an infection, such as a fever, chills, a stubborn cough or a cough that produces phlegm, persistent diarrhea, burning with urination, red or inflamed skin, or green or yellow discharge from a wound or sore.

**Progressive Multifocal Leukoencephalopathy (PML)** - Progressive multifocal leukoencephalopathy (PML) is a rare and severe viral infection of the brain that has developed in patients receiving rituximab. Some of these patients did not show signs of PML for up to 1 year after having rituximab. It is not clear whether rituximab increases the risk for PML. PML can cause brain damage, memory loss, trouble thinking, blindness, and death. Notify your study doctor immediately if you develop trouble thinking or walking, a decrease in strength in your arms or legs, or changes in your vision or hearing.

**Bowel Obstruction and Rupture** – Cancer patients treated with rituximab and chemotherapy may rarely develop blockage or rupture of the intestines. Some of these patients died. Notify your study doctor immediately if you develop pain or swelling in the stomach area or persistent vomiting.

**Decreased Blood Counts** - Rituximab may cause a decrease in the numbers of certain blood cells. This has caused patients to develop anemia (low levels of red blood cells that carry oxygen throughout your body), low numbers of platelets (the cells that help your blood clot), or low levels of white blood cells (the cells that help your body fight infections). The decrease in blood cells can last for as long as 1 year after rituximab treatment.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


**Interaction with Vaccinations** - Rituximab may interfere with your body's ability to respond to a vaccination. Certain vaccines may not be effective. Other vaccines might lead to an infection if they contain live organisms (for example, measles, mumps, rubella, or polio vaccines). Talk with your doctor before receiving any vaccinations while taking rituximab, and for 1 year after treatment has finished.

Reproductive Risks - The effects of rituximab on pregnant women, fetuses, new-born children and sperm, are unknown. If you are pregnant or breast feeding, or you are seeking to father children, you should not take this drug. If you are a woman who is able to have children, you must agree to avoid becoming pregnant while taking rituximab and for 1 year after treatment has finished (because the drug can stay in your body for a long time). Your doctor may take a sample of blood from you to test if you are pregnant before starting treatment with rituximab. If you are a man, you must agree to use contraception to prevent pregnancy while taking the drug and for twelve months thereafter. If you suspect that you, or your partner, have become pregnant, you must notify the study doctor immediately. Either of the other 2 drugs associated with this trial, bendamustine or pentostatin, may cause harm to the fetus when administered to a pregnant woman. For each of these 2 drugs, harm to the fetus has been observed in pregnant animals.

Other Effects - Other side effects that may occur during treatment with rituximab include heart failure, irregular heartbeats, and lung problems such as scarring or inflammation. If you have a history of heart problems, including irregular heartbeats, heart attacks, and/or angina (a condition where the heart doesn't receive enough blood), rituximab may worsen these conditions. Notify your study doctor immediately if you develop difficulty breathing, fainting, or pain in your chest. Immune system problems can also occur while taking rituximab. These problems can include inflammation of the eyes, nerves, blood vessels, joints, or lining of the lungs.

In addition to the effects listed above, unanticipated side effects may occur that have not been previously reported.

If you have any unusual symptoms, you should report them immediately to your doctor.

You will be kept fully informed of any events that occur during the course of the trial which might affect your safety and change your decision about continuing to participate in this trial.

Because rituximab is a mouse antibody that has been changed to make it similar to a human antibody, treatment with rituximab may cause your body to make human antibodies to the mouse-based antibody. These antibodies are called human anti-mouse antibody (HAMA) or human anti-chimeric antibody (HACA). This has happened in 1.1% (4/356) of patients and the potential response may lead to limiting the effectiveness of mouse-based antibody therapies for you in the future.

Unanticipated side effects may occur that have not been previously reported. If you have any unusual symptoms, you should report them immediately to your doctor.

# **Bendamustine toxicity**

Likely (50-60% of patients):

None

Less likely (25-50% of patients):

• Low neutrophil count

PATIENT IDENTIFICATION

## Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


# Unlikely (10-25% of patients):

- Low platelet count
- Low red blood cell count (anemia)
- Low white blood cell count
- Nausea
- Vomiting
- Fever

## Very unlikely (less than 10% of patients):

- Low blood lymphocyte count
- Diarrhea
- Fatigue
- Chills
- Allergic reaction
- Throat infection
- Other infection
- Weight loss
- High uric acid level
- Cough
- Rash
- Itching
- Liver function tests abnormalities
- Abnormal taste
- High or low blood pressure
- Fast heart rate
- Chest pain
- Itching
- Dry skin
- Abnormal blood electrolytes
- High blood sugar
- Acid reflux
- Mouth sores
- Bone pain
- Joint pain

During the intravenous infusion of bendamustine, there have been reports of drug escaping from the blood vessel into the tissues. This can cause redness, swelling, pain, infection and tissue damage.

## **Pentostatin toxicities**

## Likely (50-60% of patients):

- Nausea or vomiting
- Low white blood cell count

## PATIENT IDENTIFICATION

## Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


# Less likely (25-50% of patients):

- Fatigue
- Rash
- Low red blood cell count (anemia)
- Low platelet count
- Infection
- Fever

## Unlikely (10-25% of patients):

- Muscle aches
- Chills
- Fatigue
- Itching
- Sweating
- Diarrhea
- Decreased appetite
- Abnormal liver function tests
- Runny nose (like with allergy)
- Allergic reaction
- Infection in head or throat
- Sore throat
- Headache
- Pain
- Nerve disease
- Cough
- Lung problem
- Kidney problem

## Very unlikely (less than 10%% of patients):

- Joint pains
- Abdominal pain
- Mouth sores
- Shortness of breath
- Anxiety
- Confusion
- Insomnia
- Chest pain
- Low or high blood pressure
- Pain in abdomen
- Mouth sores
- Abnormal liver function test
- Decreased kidney function

## PATIENT IDENTIFICATION

## Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


## Risks from study procedures

#### **Blood draws**

Side effects of blood draws include pain and bruising in the area where the needle was placed, lightheadedness, and rarely, fainting and infection.

#### Risks from urine collection

There is no risk related to urine collection.

## Bone marrow biopsy and aspiration

This involves inserting a needle into a large bone such as the pelvis and removing a small amount of bone marrow fluid (aspiration) and a sample of solid bone marrow tissue (biopsy). The aspiration is usually performed first with a smaller needle than is used in the biopsy.

A numbing agent that can cause a stinging or burning sensation may be injected at the site of your bone marrow aspiration/biopsy. The needle will go through the skin into the bone and may produce a brief, sharp pain. As the sample is taken from the bone, there may be a brief, sharp pain. This procedure may cause some discomfort, however not all participants experience discomfort.

The possible side effects associated with a bone marrow aspiration/biopsy include pain, bleeding, bruising, and infection, as well as a reaction to the numbing agent. If your pain is severe or you develop a fever, please contact the study team immediately.

#### Local anesthesia

Biopsy may be done under local anesthesia. Potential side effects of local anesthesia include drowsiness, headaches, blurred vision, twitching muscles or shivering, continuing numbness, weakness or pins and needles sensation.

#### **Echocardiogram**

There is no physical risk involved with echocardiogram.

#### Electrocardiogram (EKG)

Some skin irritation can occur where the EKG electrodes are placed. Once the electrodes are placed, the test will begin, is completely painless, and generally takes less than a minute to perform. After the test, the electrodes are removed.

#### Stress test

A stress test, also called an exercise stress test, shows how your heart works during physical activity. Because exercise makes your heart pump harder and faster, an exercise stress test can reveal problems with blood flow within your heart. A stress test usually involves walking on a treadmill or riding a stationary bike your heart rhythm, blood pressure and breathing are monitored.

A stress test is generally safe, and complications are rare. Risk of complications, include:

 Low blood pressure. Blood pressure may drop during or immediately after exercise, possibly causing you to feel dizzy or faint. The problem should go away after you stop exercising.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


- Abnormal heart rhythms (arrhythmias). Arrhythmias brought on by an exercise stress test usually go away soon after you stop exercising.
- Heart attack (myocardial infarction). Although exceedingly rare, it's possible that an exercise stress test could cause a heart attack.

## **Pulmonary function tests (PFTs)**

Pulmonary function tests (PFTs) are a group of tests that measure how well your lungs work. This includes how well you're able to breathe and how effective your lungs are able to bring oxygen to the rest of your body. PFTs are usually safe for most people. However, because the test may require you to breathe in and out quickly, you may feel dizzy and there's a risk that you may faint. If you have asthma, the test may cause you to have an asthma attack. In very rare cases, PFTs may cause a collapsed lung.

#### Ultrasound

The ultrasound procedure will take about 15- 30 minutes. Ultrasound has extremely minimal risk with no use of ionizing radiation or adverse heating or pressure effects in tissue in the way that it is being utilized.

## Imaging/scans

You may receive a contrast agent injected into your arm as part of your scan. Contrast agents can cause allergic reactions and kidney damage. Allergic reactions can include mild itching associated with hives but can also result in a serious life-threatening emergency from difficulty breathing. If this occurs, it is treatable. You may feel discomfort when the contrast material is injected. You may feel warm, flushed, get a metallic taste in your mouth or, rarely, may make you vomit or feel sick to your stomach. Please ask the study doctor if you have questions about the risks of these scans.

#### Risks for MRI

Magnetic resonance imaging (MRI) uses a strong magnetic field and radio waves to take pictures of the body. We will obtain pictures of your chest, abdomen and pelvis for this study. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. People are at risk for injury from the MRI magnet if they have some kinds of metal in their body. It may be unsafe for you to have an MRI scan if you have pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metal prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, tattoos, an implanted delivery pump, or shrapnel fragments. Welders and metal workers may have small metal fragments in the eye. You will be screened for these conditions before having any MRI scan. If you have a question about metal in your body, you should inform the staff. You will be asked to complete an MRI screening form before each MRI scan you have.

In addition, all magnetic objects (like watches, coins, jewelry, and credit cards) must be removed before entering the MRI scan room.

People with fear of confined spaces may become anxious during an MRI. Those with back problems may have back pain or discomfort from lying in the scanner. The noise from the scanner is loud enough to damage hearing, especially in people who already have hearing loss. Everyone

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


having a research MRI scan will be fitted with hearing protection. If the hearing protection comes loose during the scan, you should let us know right away.

There are no known long-term risks of MRI scans.

#### Risks from Gadolinium

During part of the MRI you will receive gadolinium, a contrast agent, through an intravenous (IV) catheter (small tube). It will be done for both research and medical purposes.

It is not known if MRI with contrast is completely safe for a developing fetus. Therefore, all women of childbearing potential will have a pregnancy test performed no more than 24 hours before each MRI scan with contrast. The scan will not be done if the pregnancy test is positive.

The risks of an IV catheter include bleeding, infection, or inflammation of the skin and vein with pain and swelling.

Mild symptoms from gadolinium infusion occur in fewer than 1% of those who receive it and usually go away quickly. Mild symptoms may include coldness in the arm during the injection, a metallic taste, headache, and nausea. In an extremely small number, fewer than one in 300,000 people, more severe symptoms have been reported including shortness of breath, wheezing, hives, and lowering of blood pressure. You should not receive gadolinium if you previously had an allergic reaction to it. You will be asked about such allergic reactions before gadolinium is given.

People with kidney disease are at risk for a serious reaction to gadolinium contrast called "nephrogenic systemic fibrosis (NSF)". This condition always involves the skin and can also involve the muscles, joints, and internal organs. NSF has resulted in a very small number of deaths. A blood test of your kidney function may be done within the month before an MRI scan with gadolinium contrast. You will not receive gadolinium for a research MRI scan if your kidney function is below the safe level.

Most of the gadolinium contrast leaves the body in the urine. However, the FDA has issued a safety alert that indicates small amounts of gadolinium may remain in the body for months to years. The effects of the retained gadolinium are not clear. At this time, retained gadolinium has not been linked to health risks in people whose kidneys work well. Some types of gadolinium contrast drugs are less likely to remain in the body than others. In this study, we will use the gadolinium contrast drugs that are less likely to remain in the body.

## What are the risks of radiation from research?

During your participation in this research study, you will be exposed to radiation from up to four CT Scans. The amount of radiation exposure you will receive from these procedures is equal to approximately 5.2 rem. A rem is a unit of absorbed radiation.

Every day, people are exposed to low levels of radiation that come from the sun and the environment around them. The average person in the United States receives a radiation exposure of 0.3 rem per year from these sources. This type of radiation is called "background radiation." This study will expose you to more radiation than you get from everyday background radiation. No one knows for sure whether exposure to these low amounts of radiation is harmful to your body.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


The four CT Scans that you get in this study will expose you to the roughly the same amount of radiation as 17.3 years' worth of background radiation. Being exposed to too much radiation can cause harmful side effects such as an increase in the risk of cancer. The risk depends on how much radiation you are exposed to. Please be aware that about 40 out of 100 people (40%) will get cancer during their lifetime, and 20 out of 100 (20%) will die from cancer. The risk of getting cancer from the radiation exposure in this study is 0.5 out of 100 (0.5%) and of getting a fatal cancer is 0.3 out of 100 (0.3%).

You may not participate in this study if you are pregnant. If you are able to become pregnant, we will perform a pregnancy test before exposing you to radiation. You must tell us if you may have become pregnant within the previous 14 days because the pregnancy test is unreliable during that time.

## **Potential Benefits of Participation**

## Are there benefits to taking part in this study?

The aim of this study is to see if this combination treatment will cause improvement in your hairy cell leukemia/variant such as reduction in cancer-related symptoms. We do not know if you will receive personal medical benefit from taking part in this study. Because there is not much information about the combination of these drugs effect on your cancer, we do not know if you will benefit from taking part in this study, although the knowledge gained from this study may help us advance the understanding of the best treatment of hairy cell leukemia/variant.

## **Alternative Approaches or Treatments**

You may decide now not to receive treatment in this protocol or you may choose at any point in time to stop the drugs and withdraw from the protocol. In either case you would be returned to the care of your referring physician.

Because of the type and extent of your tumor, chemotherapy is felt to be more beneficial than surgery or radiation alone. Alternative approaches that could be used may include:

- 1. Other forms of treatment:
  - a. Several drugs can be useful in patients with HCL/HCLv, alone or in combination. These may include Cladribine, fludarabine and interferon, which are also drugs which can produce responses in HCL/HCLv, but they also can hurt the immune system.
  - b. Radiation treatment, which sometimes can control tumor growth in local areas such as lymph nodes, spleen and bones. However, this approach will not effectively treat disease that has spread beyond the areas that are irradiated.
  - c. Surgery, which can be used to remove the spleen (if this has not already been done).
- 2. Experimental agents.

#### What other choices do I have if I do not take part in this study?

Instead of being in this study, you have other options including:

- Getting treatment or care for your cancer without being in a study
- Taking part in another study

#### PATIENT IDENTIFICATION

## Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


• Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly. Instead, it tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

Please talk to your doctor about these and other options.

# **Stopping Therapy**

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest
- if your disease progresses during treatment
- if you have side effects from the treatment that your doctor thinks are too severe
- if you have another illness or medical circumstance
- if you receive radiation therapy
- if you are not following the guidelines of the study
- if you withdraw from the study

In this case, you will be informed of the reason therapy is being stopped.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. If you withdraw your consent and leave the trial, any samples of yours that have been obtained for the study and stored at the NCI can be destroyed upon request. However, any samples and data generated from the samples that have already been distributed to other researchers or placed in the research databases cannot be recalled and destroyed.

## **Conflict of Interest (COI)**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a COI Guide. You may ask your research team for a copy of the COI Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines but they do not need to report their personal finances to the NIH.

The National Institutes of Health and the research team for this study are using Rituximab (Rituxan®)developed by Genentech and Biogen IDEC through a collaboration between your study team and the companies. The companies also provide financial support for this study.

Teva Pharmaceutical Industries is providing Bendamustine (Treanda®) for this study to NIH without charge. No NIH employee involved in this study receives any payment or other benefits from Teva Pharmaceutical Industries.

**Use of Specimens and Data for Future Research** 

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


Page **14** of **18** 

To advance science, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. A researcher who wants to study the information must apply to the database and be approved. Researchers use specimens and data stored in scientific databases to advance science and learn about health and disease.

We plan to keep some of your specimens and data that we collect and use them for future research and share them with other researchers. We will not contact you to ask about each of the future uses. These specimens and data will be stripped of identifiers such as name, address or account number, so that they may be used for future research on any topic and shared broadly for research purposes. Your specimens and data will be used for research purposes only and will not benefit you. It is also possible that the stored specimens and data may never be used. Results of research done on your specimens and data will not be available to you or your doctor. It might help people who have cancer and other diseases in the future.

If you do not want your stored specimens and data used for future research, please contact us in writing and let us know that you do not want us to use your specimens and/or data. Then any specimens that have not already been used or shared will be destroyed and your data will not be used for future research. However, it may not be possible to withdraw or delete materials or data once they have been shared with other researchers.

## Samples to be saved for additional tests:

• Samples of blood or urine may be drawn to learn more about the disease hairy cell leukemia/variant, and to study the drugs used to treat this disease, including how they work to kill cancer cells, and what toxicity they might cause. You will be given the opportunity to decide whether you want to participate at the time of collection

Some of these research studies will be performed under the companion protocol 10-C-0066. You will be asked to sign another consent prior to having any samples collected.

Assays which could have an impact on both patients and their children, including studies of genetic cancer risk, will not be done.

#### COMPENSATION, REIMBURSEMENT, AND PAYMENT

# Will you receive compensation for participation in the study?

You will not receive compensation for participation in this study.

## Will you receive reimbursement or direct payment by NIH as part of your participation?

Some NIH Clinical Center studies offer reimbursement or payment for travel, lodging or meals while participating in the research. The amount, if any, is guided by NIH policies and guidelines.

On this study, the NCI will cover the cost for some of your expenses. Some of these costs may be paid directly by the NIH and some may be reimbursed after you have paid. Someone will work with you to provide more information.

## Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or related clinical care that you receive at the NIH Clinical Center.

## PATIENT IDENTIFICATION

## **Consent to Participate in a Clinical Research Study**

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


If some tests and procedures are performed outside the NIH Clinical Center, you may have to pay for these costs.

#### CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

## Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- Qualified representatives from Genentech and Biogen IDEC, the pharmaceutical company who produces rituximab, and Teva Pharmaceutical Industries, the pharmaceutical company who produces bendamustine

When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

If we share your specimens or data with other researchers, in most circumstances we will remove your identifiers before sharing your specimens or data. You should be aware that there is a slight possibility that someone could figure out the information is about you.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

### **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

## **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical records we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your medical record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

### POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

## PROBLEMS OR QUESTIONS

If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator Robert Kreitman, <u>kreitmar@mail.nih.gov</u>, 301-480-6187. You may also call the NIH Clinical Center Patient Representative at 301-496-2626, or the NIH Office of IRB Operations at 301-402-3713, if you have a research-related complaint or concern.

## CONSENT DOCUMENT

Please keep a copy of this document in case you want to read it again.

PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


IRB NUMBER: 10C0025 IRB APPROVAL DATE: 10/11/2022

| to discuss it and to ask question | ns. I consent to | o participate in this study. | |
|---|---|---|---|
| Signature of Research Particip | ant | Print Name of Research Participa | nt Date |
| about this study and have been to make research decisions on | n given the opp<br>behalf of the accable, the infor | ortunity to discuss it and to ask questic<br>dult participant unable to consent and he<br>mation in the above consent was descri- | ons. I am legally authorizate the authority to provi |
| Signature of LAR | | Print Name of LAR | Date |
| Investigator: | | | |
| Signature of Investigator | | Print Name of Investigator | Date |
| Signature of Witness | | Print Name of Witness | Date |
| NIH ADMINISTRATIVE INTERPRETER: | SECTION T | O BE COMPLETED REGARDI | NG THE USE OF A |
| the administration of informed also serve as the witness. | d consent and | speaks English and the participant's proserved as a witness. The investigator | obtaining consent may |
| the administration of informed also serve as the witness. An interpreter, or other in | d consent <u>and</u> dividual, who | | obtaining consent may a eferred language facilita ID code of the person |


CC ICF template v. 09.27.19